CLINICAL TRIAL: NCT06852183
Title: Restructuring Body Experience in Anorexia Nervosa: Virtual Reality Functionality-Focused Mirror Exposure
Acronym: VR-FME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Fatebenefratelli Hospital (Other); Centro ABA Fatebenefratelli (Unknown)
Responsible Party: Principal Investigator, Giulia Brizzi, MSC, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNR_08/2024
Record Dates: First submitted 2025-02-19; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Anorexia Nervosa
Keywords: Virtual Reality; Multisensory Integration; Anorexia Nervosa; Body Image
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Masking Description: Participants will be randomly divided into a control group (Treatment as usual - TAU) and experimental group ( TAU + Virtual Reality intervention).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-FME (Experimental): The VR-FME protocol integrates multiple therapeutic approaches within an immersive virtual environment. Each 60-minute session begins with embodiment induction, where participants experience synchronized multisensory stimulation to create embodiment over their virtual body. Then, various therapeutic techniques - including cognitive dissonance mirror exposure, functionality-focused mirror exposure, and compassionate body scan exercises - will be used. Each of the 8 sessions will work on a specific aspect to address different levels of body image disturbance. The intervention structure begins with an initial assessment and familiarization phase in Week 1, followed by intensive body-focused work in Weeks 2-4.
  Interventions: Other: VR -FME
- TAU (Active Comparator): For the entire duration of the protocol, both the experimental group (VR-FME) and the control groups will carry out the standard intervention protocol proposed by the treatment center, which consists of an outpatient program that includes weekly internal-nutritional visits, psychotherapy and NPIA assessments to also monitor the pharmacological therapy. Therefore, if the experimental group carries out the standard procedure (Treatment As Usual - TAU) in addition to the VR body image protocol (VR-FME + TAU), the control group will be subjected to the standard treatment path (TAU).
  Interventions: Other: VR -FME

INTERVENTIONS:
Other: VR -FME — The VR-FME intervention specifically focuses on improving body representation and the body-self relationship by working on multisensory integration processes and embodied cognition techniques. This is thanks to the combination of immersive virtual reality experiences of body illusion combined with traditional psychological techniques. The experimental group will receive this intervention in addition to the usual treatment, which will continue as usual for the control group. The intervention consists of 8 sessions spread over 4 weeks, with 2 sessions per week.

SUMMARY:
Background: Body image disturbance remains a core therapeutic challenge in Anorexia Nervosa (AN) treatment, necessitating innovative intervention approaches. This study protocol describes a randomized controlled trial investigating Virtual Reality Functionality-Focused Mirror Exposure (VR-FME), a novel intervention targeting the perceptual, affective, and cognitive dimensions of body image disturbance in AN patients.

Methods: This single-blind, parallel-group randomized controlled trial will evaluate the efficacy of VR-FME as an adjunct to treatment as usual (TAU). Participants with AN will be randomly allocated to receive either VR-FME combined with TAU or TAU alone. The intervention specifically addresses altered body image through immersive virtual reality technology, providing controlled exposure and cognitive restructuring opportunities.

Primary Outcome: The primary outcome measure will assess changes in body image disturbance severity and core eating disorder symptomatology. We hypothesize that the integration of VR-FME with TAU will demonstrate superior therapeutic outcomes compared to TAU alone.

Significance: This protocol represents an innovative approach to addressing body image disturbance in AN, potentially enhancing current therapeutic strategies through the integration of immersive virtual reality technology. The findings will contribute to the evolving landscape of technology-enhanced interventions for eating disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age: between 16-24.
* Primary diagnosis of Anorexia Nervosa
* BMI > 14.5
* No current diagnosis or previous diagnosis for neurological disorders
* Females
* Fluency in Italian
* Ability to provide informed consent (and parental consent for minors)

Exclusion Criteria:

* Anorexia Nervosa is not a primary diagnosis
* Age < 16
* BMI < 14.5
* Conditions that could interfere with VR use (e.g., neurological conditions, severe visual impairments, vestibular disorders)
* Males
* Substance abuse, active suicidal ideation, severe psychiatric comorbidities
* Pregrancy
* Ongoing participation in other clinical trials
* Inability to commit to the full duration of the study

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Eating Disorder Inventory 3 | Before the intervention, after the end of the intervention (at the end of the 4th week) and after one month after the intervention ended
  Eating Disorder Inventory 3 (EDI-3): The EDI-3 is a widely used self-report and standardized measure to assess symptomatology and psychological features relevant to developing and maintaining EDs. The third version (EDI-3) includes 91 items classified into 12 scales, with a six-point Likert scale for each answer ranging from 0 (never) to 5 (always).
Physical Appearance State and Trait Anxiety Scale | Before the intervention, after the end of the intervention (at the end of the 4th week) and after one month after the intervention ended
  Physical Appearance State and Trait Anxiety Scale (PASTAS): The PASTAS is a reliable and valid measure for the assessment of trait and state body image anxiety. Patients had to rate, on a five-point scale ranging from 0 (never) to 5 (always), if they felt anxious or nervous about their physical appearance, including any tension, negative thoughts, and physiological responses. This tool has been previously used in research studies including Italian samples.
Body Mass Index | Before the intervention, after the end of the intervention (at the end of the 4th week) and after one month after the intervention ended
  Body Mass Index (BMI)
Body Image Assessment Scale - Body Dimensions | Before the intervention, after the end of the intervention (at the end of the 4th week) and after one month after the intervention ended
  The Body Image Assessment Scale-Body Dimensions (BIAS-BD): The BIAS-BD is used to assess the perceptual and emotional components of BIDs. This test assesses the discrepancy between the perceived body size and the self-determined ideal body size (to measure body dissatisfaction). Furthermore, it also reveals the discrepancy between the perceived body size and the real body size (to measure body distortion). The scale presents a range of 17 silhouettes, with different versions for women and me
Body Size Estimation Task | Before the intervention, after the end of the intervention (at the end of the 4th week) and after one month after the intervention ended
  Body Size Estimation Task (BES): it is a behavioral task in which participants are asked to estimate the measure of specific body parts (i.e., shoulders, hips, and waist).
Body Appreciation Scale-2 | Before the intervention, after the end of the intervention (at the end of the 4th week) and after one month after the intervention ended
  Body Appreciation Scale-2 (BAS-2): The BAS-2 is a 10-item measure assessing body appreciation. Participants rate statements on Likert-type scales from 1 (never) to 5 (always). Items are averaged; higher scores indicate greater body appreciation. Example items include: "I respect my body"; "I take a positive attitude towards my body"; and "I am comfortable in my body". This tool has been validated in Italian.
Objectified Body Consciousness Scale | Before the intervention, after the end of the intervention (at the end of the 4th week) and after one month after the intervention ended
  Objectified Body Consciousness Scale (OBCS): The OBCS contains 24 items grouped into three subscales: body surveillance, body shame, and appearance control beliefs. Each subscale contains eight items, rated on a 7- 7-point Likert-type scale (1 =strongly disagree, 7 = strongly agree). Subscale items are averaged and higher scores indicate a greater manifestation of the particular variable measured. This tool has been validated in Italian.
Body Uneasiness Test | Before the intervention, after the end of the intervention (at the end of the 4th week) and after one month after the intervention ended
  Body Uneasiness Test (BUT): The BUT is a 34-item self-report questionnaire focusing on body dissatisfaction and body-related emotions such as anxiety, alarm, and embarrassment. It is composed of five subscales - weight phobia, body image concern, avoidance, compulsive self-monitoring, depersonalization - and a general score. This tool has been validated in Italian.

SECONDARY OUTCOMES:
Qualitative feedback survey | After the end of the intervention (week 4)
  Qualitative feedback from participants

IPD SHARING:
Plan to Share IPD: Yes